CLINICAL TRIAL: NCT03616210
Title: Protective Versus Conventional Mechanical Ventilation for Peripheral Vascular Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 61485616.0.0000.5327
Record Dates: First submitted 2018-04-26; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Lung Diseases
Keywords: mechanical ventilation; protective ventilation; vascular surgery; postoperative pulmonary complications
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protective ventilation (Experimental): Protective ventilation strategy (tidal volume of 6 to 7 ml.kg-1 of predicted body weight and PEEP of 6 to 8 cmH2O)
  Interventions: Procedure: Protective ventilation
- Conventional ventilation (No Intervention): Conventional mechanical ventilation (tidal volume between 9 to 10 ml.kg-1 of predicted body weight and PEEP between 3 and 5 cmH2O)

INTERVENTIONS:
Procedure: Protective ventilation — Protective ventilation strategy with tidal volume of 6 to 7 ml.kg-1 of predicted body weight and PEEP of 6 to 8 cmH2O.
  Arms: Protective ventilation

SUMMARY:
Background and goal of the study: Postoperative complications following major surgeries are associated with a significant increase in costs and mortality. There is increasing evidence that mechanical ventilation with a protective strategy using low tidal volume prevents postoperative pulmonary complications. Peripheral vascular surgeries include particularly surgeries for arterial revascularization of the lower limbs in patients with advanced peripheral vascular disease. These procedures are strongly associated with major cardiovascular morbidity postoperatively. In this specific group of patients, the presence of postoperative pulmonary complications (PPC) may be associated with worsening of clinical outcomes with a consequent significant increase in perioperative morbidity.

Subjects and methods: In this study, the investigators aimed to compare the effects of controlled mechanical ventilation with the use of a protective strategy (low tidal volume associated with elevated PEEP) when compared to the conventional strategy (higher tidal volume associated with reduced PEEP levels) on the rate of PPC in patients undergoing peripheral vascular surgery. This study was delineated as a prospective trial, compared to the control group (conventional ventilation strategy). Patients and researchers were blinded during data collection. The investigators included adult patients, ASA status II to IV, aged over 18 years, scheduled to undergo lower limb arterial bypass surgery. Patients were randomized to treatment with conventional mechanical ventilation (tidal volume between 9 to 10 ml.kg-1 of predicted body weight and PEEP between 3 and 5 cmH2O - Group I or control) or treatment with protective ventilation strategy (tidal volume of 6 to 7 ml.kg-1 of predicted body weight and PEEP of 6 to 8 cmH2O - Group II or treatment). The primary outcome was PPC and the secondary endpoint included hemodynamic and metabolic changes perioperatively. Statistical analysis was performed using the intention-to-treat method.

ELIGIBILITY:
Inclusion Criteria:

* This study enrolled only patients displaying peripheral occlusive arterial disease and scheduled to undergo an elective peripheral artery bypass surgery.

Exclusion Criteria:

* The illiterate or who do not understand Portuguese language, those who had a body-mass index (BMI) higher than 35 kg/m2, had severe pulmonary comorbidities or another disorder that might compromise a safe trial procedure and those who refused to participate of the study or who had already participated in other studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | 7 days
  The main outcome was the presence of any pulmonary complication (composite endpoint) after surgery and until discharge. These pulmonary complications included severe hypoxemia, suspected pulmonary infection, documented atelectasis or pulmonary infiltrate, bronchospasm, pulmonary edema, pleural effusion, pneumothorax, or development of ARDS. The presence of at least one of the findings described above was considered as a positive primary outcome.

SECONDARY OUTCOMES:
Perioperative hemodynamic complications | 7 days
  Hypotension and need for continuous vasopressors (i.e., systolic arterial blood pressure < 90 mmHg for more than 5 min).

CONTACTS AND LOCATIONS:
Overall Officials: Andre P Schmidt, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Andre P Schmidt, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No